CLINICAL TRIAL: NCT01534091
Title: Enhancing the Amount of Physical Activity Carried Out by Overweight Children at Leisure Time
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of cooperation by the participants
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MeirMc02711CTIL
Record Dates: First submitted 2012-01-18; First posted 2012-02-16 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2013-10

CONDITIONS: Obesity
Keywords: overweight; obese; children; exercise; physical activity; pedometer
MeSH Terms: conditions — Obesity; Overweight; Motor Activity | interventions — Organization and Administration; Exercise; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pedometer with supervision (Active Comparator): Participants will get pedometers to evaluate their daily PA. The sport center stuff will review the child weekly reports, guide the child, encourage him and supervise that the recommended PA level is achieved.
  Interventions: Behavioral: Pedometer with supervision
- Pedometer without supervision (Active Comparator): Participants will get pedometers to evaluate their daily PA. The sport center stuff won't give any recommendation or supervision for PA level.
  Interventions: Behavioral: Pedometer without supervision
- Control group (No Intervention): Overweight & obese children not participating in an intervention.

INTERVENTIONS:
Behavioral: Pedometer with supervision
  Other Names: exercise + diet + pedometer
  Arms: Pedometer with supervision
Behavioral: Pedometer without supervision
  Other Names: exercise + diet + closed pedometer
  Arms: Pedometer without supervision

SUMMARY:
The purpose of this study is to examine if internet supervised by pedometer will contribute to enhance the amount of physical activity at leisure time by obese children.

The investigators hypothesize that using pedometer will increase the amount of physical activity done by obese children in the afternoon and will improve the likelihood of success in the intervention program.

DETAILED DESCRIPTION:
Childhood overweight & obesity is the most common chronic disease in the western society. The prevalence of childhood obesity in Israel is among the highest in Europe. Recent data suggest that the recommended treatment for childhood obesity should be intense, multi-disciplinary intervention, including dietary, behavioral and physical activity components. Such a program exists at the Meir Medical Center in Israel for a few years with promising results.

The program includes: physical activity(PA)exercise (twice a week/1h), dietary guidance, medical supervision and behavioral intervention. The participants are asked to enhance PA at their leisure time, and to report to their coaches. Yet, the amount of time they actually exercise is not controled by us.

This study will include 3 groups of overweight& obese children:

1. Intervention with pedometers and supervision.
2. Intervention with pedometer without supervision.
3. Control. Obese and overweight children not taking part in a treatment program.

ELIGIBILITY:
Inclusion Criteria:

* overweight/obese children
* age 5-18
* boys and girls

Exclusion Criteria:

* children with genetic obesity or obesity cased by a disease

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2012-05; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Decline in BMI percentiles | 3 months
  BMI percentiles will be calculated at the beginning and in the end of the study

SECONDARY OUTCOMES:
Aerobic fitness | 3 months intervention
  15 minutes of running or walking test

CONTACTS AND LOCATIONS:
Overall Officials: Dan Nemet, Prof. MD, Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel